CLINICAL TRIAL: NCT05638841
Title: Prospective Cohort Study of the Risk of Recurrent Atrial Fibrillation After Radiofrequency Ablation
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-653-01
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- atrial fibrillation: After radiofrequency ablation of patients with atrial fibrillation
  Interventions: Other: After radiofrequency ablation of atrial fibrillation

INTERVENTIONS:
Other: After radiofrequency ablation of atrial fibrillation — This study imposed an intervention. Clinical data were obtained by telephone or outpatient follow-up.

SUMMARY:
In this study, the continuous inclusion of atrial fibrillation patients treated by catheter ablation in the Department of Cardiology, Peking University Third Hospital, through the collection of clinical data and outpatient follow-up, to explore the risk factors of atrial fibrillation recurrence after catheter ablation and the influencing factors of major clinical events in atrial fibrillation patients, and further guide the management mode of atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age > 18
* 2) ECG or holter electrocardiogram confirmed atrial fibrillation

Exclusion Criteria:

* 1) Hematological diseases, autoimmune diseases and malignant tumors
* 2) Immobility caused by hemiplegia or severe trauma
* 3) The expected survival time is less than 2 years
* 4) Poor compliance and high risk of expected loss of follow-up
* 5) Disorders of consciousness or Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, atrial fibrillation patients who meet the inclusion criteria and those who do not meet the exclusion criteria were admitted to the Department of Cardiology of Peking University Third Hospital after catheter ablation from December 31, 2022 to December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compound cardiovascular event | 24 months
  Stroke, hemorrhage, re-hospitalization for atrial fibrillation and heart failure, and all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking-University-Third-Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No